CLINICAL TRIAL: NCT00879424
Title: Randomized Trial of Vitamin D Supplementation in Winter-related, Childhood Atopic Dermatitis
Brief Title: Vitamin D Supplementation in Childhood Atopic Dermatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Carlos A. Camargo, Jr., Physician, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CeDAR-01
Record Dates: First submitted 2009-04-09; First posted 2009-04-10 (Estimated); Last update posted 2016-12-22 (Estimated); Status verified 2016-12

CONDITIONS: Atopic Dermatitis
Keywords: vitamin D; atopic dermatitis; eczema; winter
MeSH Terms: conditions — Dermatitis, Atopic; Eczema | interventions — Cholecalciferol; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Dietary Supplement: cholecalciferol (vitamin D)
- 2 (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: cholecalciferol (vitamin D) — 1000 IU once daily x 1 month
  Experimental group will receive Ddrops (Toronto, Canada). Placebo group will receive placebo drops.
  Other Names: Experimental group will receive Ddrops (Toronto, Canada).; Placebo group will receive placebo drops.
  Arms: 1
Dietary Supplement: Placebo — 1000 IU once daily x 1 month
  Experimental group will receive Ddrops (Toronto, Canada). Placebo group will receive placebo drops.
  Arms: 2

SUMMARY:
The goal of this clinical trial is to investigate the therapeutic role of vitamin D supplementation in a subset of patients with atopic dermatitis (AD): children with disease onset or worsening in the winter. The investigators hypothesis is that (1) vitamin D supplementation in patients with either wintertime onset or exacerbation of AD will improve Eczema Area and Severity Index (EASI) scores, and (2) vitamin D supplementation will improve the Investigator's Global Assessment.

ELIGIBILITY:
Inclusion Criteria:

* Age 2-17 years
* AD rated 10-72 by EASI scale
* Wintertime onset or exacerbation of AD

Exclusion Criteria:

* Active skin infection
* History of summertime onset or exacerbation of AD
* History of underlying illness causing immunosuppression within the past 2 years (eg. hematologic malignancies)
* Medications causing iatrogenic immunosuppression (eg. cyclosporine; azathioprine, oral steroids) taken within the past month
* Parathyroid disease
* Acute or chronic renal disease
* Hypercalcemia or hypocalcemia
* Thyroid disease
* History of osteomalacia or Paget's disease of bone
* History of malabsorption (eg cystic fibrosis)
* Planned trip to sunny climate during the one-month study

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 107 (Actual)
Dates: Start 2009-02; Primary Completion 2009-04 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
EASI score | 1 month
Investigator Global Assessment (IGA) | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Carlos A. Camargo, MD, DrPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- National Dermatology Center, Ulaanbaatar, Mongolia

REFERENCES:
- [Background] Sidbury R, Sullivan AF, Thadhani RI, Camargo CA Jr. Randomized controlled trial of vitamin D supplementation for winter-related atopic dermatitis in Boston: a pilot study. Br J Dermatol. 2008 Jul;159(1):245-7. doi: 10.1111/j.1365-2133.2008.08601.x. Epub 2008 Jul 1. No abstract available. PMID 18489598
- [Result] Camargo CA Jr, Ganmaa D, Sidbury R, Erdenedelger Kh, Radnaakhand N, Khandsuren B. Randomized trial of vitamin D supplementation for winter-related atopic dermatitis in children. J Allergy Clin Immunol. 2014 Oct;134(4):831-835.e1. doi: 10.1016/j.jaci.2014.08.002. PMID 25282565
- [Derived] Huey SL, Acharya N, Silver A, Sheni R, Yu EA, Pena-Rosas JP, Mehta S. Effects of oral vitamin D supplementation on linear growth and other health outcomes among children under five years of age. Cochrane Database Syst Rev. 2020 Dec 8;12(12):CD012875. doi: 10.1002/14651858.CD012875.pub2. PMID 33305842